CLINICAL TRIAL: NCT04676776
Title: Assessing Use Of Mifepristone After Progestin Priming For Use As "Missed Period Pills"
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gynuity Health Projects (Other)
Collaborators: Cuidado Integral de la Mujer, Gineclinic, S.C. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 8005
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Missed Menstrual Period
MeSH Terms: interventions — Levonorgestrel; Mifepristone

STUDY DESIGN:
Intervention Model Description: Simon's two-stage design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Missed period pill regimen (Experimental): 1.5 mg levonorgestrel given on day 1 200 mg mifepristone given on day 3
  Interventions: Drug: Levonorgestrel; Drug: Mifepristone

INTERVENTIONS:
Drug: Levonorgestrel — All participants receive 1.5 mg levonorgestrel on day 1
Drug: Mifepristone — All participants receive 200 mg mifepristone on day 3

SUMMARY:
This study will assess the effectiveness and acceptability of a 3-day missed period pill regimen.

DETAILED DESCRIPTION:
Missed period pills (MPPs) are medications used for uterine evacuation among women with late menses who have not confirmed pregnancy status. Provision of MPPs could expand reproductive service options for individuals in a variety of settings. This study will collect data on the efficacy, safety, and acceptability of a 3-day missed period pill regimen among individuals with missed menses of 1-10 days

ELIGIBILITY:
Inclusion Criteria:

* Age 18-49 years
* General good health
* Does not want to be pregnant
* History of regular monthly menstrual cycles (±3 days)
* Missed menses of 1 to 10 days as verified by report of last menstrual period
* Sexual activity in the past month
* Willing and able to sign consent forms
* Willing to return for a follow-up visit
* Willing to provide a urine sample at enrollment and at follow-up

Exclusion Criteria:

* Known allergies or contraindications to mifepristone
* Symptoms of or risk factors for ectopic pregnancy, such as vaginal bleeding or spotting within the past week; unilateral pelvic pain or significant bilateral pelvic pain within the past week; prior ectopic pregnancy; prior permanent contraception or other tubal surgery
* Current use of an IUD, contraceptive implant or injectable

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 139 (Estimated)
Dates: Start 2021-01-25 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of missed period pill regimen | Up to 28 days after administration of levonorgestrel
  Proportion of participants not pregnant at follow-up among those who were pregnant at enrollment

SECONDARY OUTCOMES:
Effectiveness of missed period pill regimen | Up to 28 days after administration of levonorgestrel
  Proportion of all enrolled participants not pregnant at follow-up (among those who were and were not pregnant at enrollment)
Effectiveness at inducing return of menses within 10 days | Up to 10 days after administration of levonorgestrel
  Proportion of participants reporting return of missed menses within 10 days of initiating missed period pill regimen
Occurrence of treatment-emergent adverse events and/or side effects (safety and tolerability) | Up to 28 days after administration of levonorgestrel
  Proportion of participants who report adverse events and/or side effects
Acceptability of missed period pills | Up to 28 days after administration of levonorgestrel
  Proportion of participants who report that the missed period pill service was acceptable or highly acceptable to them

CONTACTS AND LOCATIONS:
Overall Officials: Beverly H Winikoff, MD, Principal Investigator — Gynuity Health Projects; Holly A Anger, Study Director — Gynuity Health Projects
Locations (1):
- Cuidado Integral de la Mujer, Gineclinic, S.C, Mexico City, Mexico